CLINICAL TRIAL: NCT07218926
Title: A Phase 3, Randomized, Multicenter, Open-Label Study of IDRX-42 (GSK6042981) Versus Sunitinib in Participants With Metastatic and/or Unresectable Gastrointestinal Stromal Tumors (GIST) After Imatinib Therapy (StrateGIST 3)
Brief Title: A Study of IDRX-42 (GSK6042981) Versus (vs) Sunitinib in Participants With Gastrointestinal Stromal Tumors After Imatinib Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300383; 2025-522229-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Neoplasms
Keywords: GSK6042981; IDRX-42; Sunitinib; Imatinib; Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Neoplasms; Gastrointestinal Stromal Tumors | interventions — IDRX-42; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDRX-42 (GSK6042981) (Experimental)
  Interventions: Drug: IDRX-42
- Sunitinib (Active Comparator)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: IDRX-42 — IDRX-42 will be administered.
  Other Names: GSK6042981
  Arms: IDRX-42 (GSK6042981)
Drug: Sunitinib — Sunitinib will be administered.
  Arms: Sunitinib

SUMMARY:
The purpose of this study is to find out if a new drug, called IDRX-42 (also known as GSK6042981), is effective in treating adults with a type of cancer called Gastrointestinal Stromal Tumors (GIST) when compared to another drug named sunitinib. The study will see if IDRX-42 works well and is safe for participants whose GIST has spread or cannot be surgically removed, and who have already taken the drug imatinib.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed GIST that is metastatic and/or surgically unresectable.
* Documented disease progression on or intolerance to imatinib administered for first-line treatment of unresectable/metastatic disease.
* Tumor tissue must be available to be submitted to the central laboratory for retrospective biomarker analysis. The sample may be from archival tissue or a new biopsy. Tissue samples are not required to be submitted centrally prior to randomization.

Exclusion Criteria:

* Known untreated or active central nervous system metastases.
* Participants with a known allergy or hypersensitivity to any component of IDRX-42 (GSK6042981) or sunitinib. Participants with a history of Stevens-Johnson syndrome on a prior Tyrosine kinase inhibitor (TKI) are excluded.
* Has a malignancy (except disease under study) that has progressed or required active treatment within the past 24 months except for basal cell or squamous cell carcinomas of the skin or in-situ carcinomas [e.g., breast, cervix, bladder] that have been resected with no evidence of metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2030-11-29 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 130 weeks
  PFS is defined as time from the date of randomization to the date of disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 261 weeks
  OS is defined as time from the date of randomization to the date of death due to any cause.
Progression-Free Survival (PFS) | Up to approximately 261 weeks
  PFS is defined as time from the date of randomization to the date of disease progression or death due to any cause, whichever occurs first.
Confirmed Overall Objective Response Rate (ORR) | Up to approximately 261 weeks
  ORR is defined as the percentage of participants with the best overall confirmed partial response (PR) or better.
Time to Response (TTR) | Up to approximately 261 weeks
  TTR is defined as time from randomization until the first documented PR or complete response (CR) that will be subsequently confirmed.
Time from initial study randomization to second disease progression or death after starting the next line of treatment (PFS2) | Up to approximately 261 weeks
  PFS2 is defined as the time from initial study randomization to second disease progression or death after starting the next line of treatment.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core Module (EORTC QLQ-C30) | Baseline (Day 1) and up to approximately 261 weeks
  The EORTC QLQ-C30 includes 30-item questionnaire for evaluating the health-related quality of life (HRQoL) of participants participating in cancer clinical studies. These include functional scales, symptom scales, global health status scale, and single item scales. Scores are averaged and transformed to 0 to 100. Higher scores indicate greater functioning, better global health status, or more severe symptoms
Time To Confirmed Deterioration (TTCD) | Up to approximately 261 weeks
  TTCD is defined as the time from the date of randomization to the first confirmed clinically meaningful deterioration based on the EORTC QLQ-C30.
Plasma concentrations of IDRX-42 (GSK6042981) | Up to approximately 261 weeks
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to approximately 261 weeks
Number of Participants with TEAEs and SAEs by severity | Up to approximately 261 weeks
Number of Participants with dose reductions, interruptions and discontinuation of study treatment due to toxicity | Up to approximately 261 weeks
Number of participants with symptomatic adverse events (AEs), by severity, as measured by the Patient-reported outcome Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to approximately 261 weeks
  The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicities in participants in cancer clinical trials. The PRO-CTCAE includes an item library of 124 items representing 78 symptomatic toxicities drawn from the CTCAE.
Number of participants with bothersome AEs/tolerability as measured by the Functional Assessment of Cancer Therapy - General (FACT-GP5) | Up to approximately 261 weeks
  The FACT GP5 is an assessment focused on the overall side effects impact to inform the tolerability of a treatment. The FACT GP5 ("I am bothered by side effects of treatment") responses are given on a 5-point Likert type scale. The response scale ranges from 0 (Not at all) to 4 (Very much). Higher scores indicate a higher degree of AE bother.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (7):
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Tacoma, Washington
- GSK Investigational Site, Toronto, Ontario, Canada
- Japan (7):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Taiwan (3):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.